CLINICAL TRIAL: NCT06553209
Title: A Randomized, Double-blind, Single/Multiple Dose Escalation, Placebo-controlled Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM512 in Healthy Subjects and Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Study of CM512 in Healthy Subjects and Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM512-100001
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 2 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 3 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 4 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 5 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 6 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo
- Group 7 (Experimental)
  Interventions: Biological: CM512; Drug: Placebo

INTERVENTIONS:
Biological: CM512 — CM512 injection
Drug: Placebo — Placebo

SUMMARY:
This is a randomized, double-blind, single/multiple dose escalation, placebo-controlled phase I study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of CM512 in healthy subjects and patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written informed consent form (ICF).
* Body mass index (BMI) ranges from 18.0 to 26.0 kg/m2 (including boundary values).

Exclusion Criteria:

* Have participated in any clinical trials of drugs or medical devices within 3 months before the screening.
* Have severe infections, severe injuries, or undergone major surgical procedures within 3 months before screening.
* Have lost more than 400 mL of blood due to blood donation or other reasons within 3 months before screening.
* Positive drug abuse test or positive alcohol breath test result.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 141 days or up to 169 days
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Li, Principal Investigator — West China Hospital; Ping Feng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No